CLINICAL TRIAL: NCT05496959
Title: 177-Lutetium-PSMA Neoadjuvant to Ablative Radiotherapy for Oligorecurrent Prostate Cancer (Lunar)
Brief Title: 177-Lutetium-PSMA Before Stereotactic Body Radiotherapy for the Treatment of Oligorecurrent Prostate Cancer, The LUNAR Study
Acronym: LUNAR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-000750; NCI-2022-05748 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Oligometastatic Prostate Carcinoma; Prostate Adenocarcinoma; Recurrent Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (SBRT) (Active Comparator): Beginning on day 1, patients undergo SBRT to all lesions for 1, 3, or 5 treatment doses (fractions) over the span of 10-20 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Radiation: Stereotactic Body Radiation Therapy
- Arm 2 (177Lu-PNT2002, SBRT) (Experimental): Patients receive 177Lu-PNT2002 IV over 1-10 minutes on days -112 and -56 in the absence of disease progression or unacceptable toxicity. Beginning on day 1, patients then undergo SBRT to all lesions for 1, 3, or 5 treatment doses (fractions) over the span of 10-20 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lutetium Lu-177 PNT2002; Other: Quality-of-Life Assessment; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Lutetium Lu-177 PNT2002 — Given IV
  Other Names: 177Lu-labeled PNT2002; 177Lu-PNT2002; [Lu-177]-PNT2002; [Lu-177]-PSMA-I and T; Lu177-PNT2002; Lutetium Lu-177-PNT2002
  Arms: Arm 2 (177Lu-PNT2002, SBRT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial tests whether 177-Lutetium-PSMA given before stereotactic body radiotherapy (SBRT) works to improve cancer control rate in patients with 1-5 prostate cancer tumors that have come back after prior treatment (oligorecurrent). Radioactive drugs, such as 177-Lutetium-PSMA, may carry radiation directly to tumor cells and not harm normal cells. SBRT uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving 177-Lutetium-PSMA before SBRT may make the SBRT more effective.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess progression-free survival for men with oligorecurrent prostate cancer after stereotactic body radiotherapy (SBRT) versus SBRT plus neoadjuvant lutetium Lu-177 PNT2002 (177Lu-PNT2002), with progression defined on the basis of prostate-specific membrane antigen positron emission tomography/computerized tomography (PSMA PET/CT) scans obtained at standard intervals (12 months and 24 months post-SBRT) or at the time of prostate-specific antigen (PSA)-based biochemical progression, or initiation of salvage therapy or death.

SECONDARY OBJECTIVES:

I. To evaluate disease burden of disease (including local control of irradiated lesions and presence of other disease) on a PSMA PET/CT obtained 24 months after SBRT of SBRT versus SBRT + 177Lu-PNT2002 in patients with oligometastatic disease who have not progressed by that point.

II. To assess physician-scored toxicity (Common Terminology Criteria for Adverse Events version 5.0 [CTCAE v 5.0]) of SBRT versus SBRT + 177Lu-PNT2002 in patients with oligometastatic disease.

III. To assess patient-reported quality of life (based on the brief pain inventory scale) after SBRT versus SBRT + 177Lu-PNT2002 in patients with oligometastatic disease.

IV. To assess androgen deprivation therapy (ADT)-free survival after SBRT versus SBRT + 177Lu-PNT2002 in patients with oligometastatic disease.

V. To determine local control of irradiated lesion at 12 months after SBRT versus SBRT + 177Lu-PNT2002 in patients with oligometastatic disease (based on a scheduled PSMA-PET).

VI. To assess time to locoregional progression, time to distant progression, time to new metastasis, and duration of response after SBRT versus SBRT + 177Lu-PNT2002 in patients with oligometastatic disease (based on standard of care imaging).

CORRELATIVE OBJECTIVES:

I. To enumerate circulating tumor cells (CTCs) and circulating tumor deoxyribonucleic acid (ctDNA) at baseline, 3 months, 6 months, and 12 months after SBRT.

II. To quantitatively sequence T-cell receptor (TCR) repertoires using peripheral blood monocytes at baseline, 3 months, 6 months, and 12 months after SBRT.

III. To perform radiomics analysis on PSMA PET/CT scans performed at +12 months (mo.), +24 months post-SBRT, or at time of progression.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Beginning on day 1, patients undergo SBRT to all lesions for 1, 3, or 5 treatment doses (fractions) over the span of 10-20 days in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive 177Lu-PNT2002 intravenously (IV) over 1-10 minutes on days -112 and -56 in the absence of disease progression or unacceptable toxicity. Beginning on day 1, patients then undergo SBRT to all lesions for 1, 3, or 5 treatment doses (fractions) over the span of 10-20 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment patients are followed up at 1, 3, 6, 9, and 12 months, then every 6 months until 60 months of total follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Oligorecurrent prostate cancer as determined by the presence of 1-5 asymptomatic lesions outside the prostate or prostate bed identified on PSMA PET/CT by local readers
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* No indication for urgent or emergent radiation
* Histologic confirmation of prostate adenocarcinoma (histology from original treatment acceptable)
* White blood cell count >= 2.5 × 10^9/L
* Platelets >= 100 × 10^9/L
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 × institutional upper limit of normal (ULN); or up to 3 × ULN if known history of Gilbert's syndrome
* Alanine aminotransferase or aspartate aminotransferase =< 3.0 × ULN or =< 5.0 × ULN for patients with liver metastases
* Serum creatinine =< 1.5 × ULN or creatinine clearance >= 50 mL/min
* Serum albumin > 3.0 g/dL
* Partner and patient must use a method of birth control with adequate barrier protection, deemed acceptable by the principal investigator during the study and for 3 months after last study drug administration
* Ability to understand, and willingness to sign, the written informed consent

Exclusion Criteria:

* Patients with neuroendocrine or small cell carcinoma of the prostate
* Patients with castrate-resistant disease (i.e., PSA > 0.5 ng/mL with serum testosterone < 150 ng/dL)
* Patients who received androgen deprivation therapy within 6 months of trial enrollment
* Concurrent systemic therapy for a solid organ malignancy
* Spinal cord compression
* Inability to lie flat
* Known hypersensitivity to components of 177Lu-PNT2002
* Serum creatinine > 1.5 × ULN or creatinine clearance < 50 mL/min
* Total bilirubin > 1.5 × ULN or > 3.0 × ULN if known history of Gilbert's syndrome
* Alanine aminotransferase or aspartate aminotransferase > 3 × ULN (or 5 × ULN for patients with known liver metastases)
* De novo oligometastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2032-09-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
Prostate-specific membrane antigen positron emission tomography/computerized tomography (PSMA PET/CT)-based progression-free survival (PFS) | Time from the date of stereotactic body radiotherapy (SBRT) completion to the date of disease progression or death, whichever happens earlier, assessed up to 24 months
  Will compare PSMA PET/CT-based PFS for patients with oligoprogressive prostate cancer treated with SBRT to all known sites of disease on PSMA PET/CT versus patients treated with 177Lu-PNT2002 prior to SBRT to all known sites of disease. PSMA PET/CT-based progression is defined as either (a) a new lesion on PSMA PET/CT with or without a serum prostate-specific antigen (PSA) increase or (b) local progression on PSMA (> 30% increase in lesion standard uptake value [SUV] or increase of > 20% in the sum of the longest diameter of all target lesions), regardless of new lesions, and a serum PSA increase. A serum PSA increase for the purposes of this definition will be based on the definition of PSA-based progression. The Kaplan-Meier (KM) method will be used to summarize PFS and log-rank test will be used to compare PFS between the two arms.

SECONDARY OUTCOMES:
Disease progression | At 24 months
  Progression as based PSMA PET/CT scan (with progression). Will be analyzed descriptively.
PSA-based progression | Up to 24 months
  Defined as follows: (a) For pre-enrollment PSA < 0.5 ng/mL, PSA-based progression defined as 0.2 ng/mL increase and (b) For pre-enrollment PSA >= 0.5 ng/mL, PSA-based progression defined as 50% increase over pre-treatment value.
Incidence of adverse events (AEs) | Up to 60 months
  Acute and late physician-scored toxicity Common Terminology Criteria for Adverse Events (CTCAE version 5.0 scale). AEs will be summarized by type and grade. All patients who receive at least one fraction of SBRT in the control arm will be evaluable for toxicity from the time of their first treatment from SBRT; all patients who receive 177Lu-PNT2002 in the experimental arm will be evaluable for toxicity from the time of their first treatment with 177Lu-PNT2002.
Patient-reported quality of life as reported by the Brief Pain Inventory form | Baseline up to 1 year
  Quality of life following SBRT versus 177Lu-PNT2002 +SBRT will be evaluated based on responses to the Brief Pain Inventory form, which will be tabulated at baseline and each follow-up visit (3 months, 6 months, 9 months and 1 year).
  The Brief Pain Inventory is a self-administered 9-item questionnaire, tabular scored from 0 - 130 with lower scores indicating a better outcome.
Androgen deprivation therapy-free survival (ADT-FS) | Time from starting treatment to the time of initiation of palliative ADT, assessed up to 60 months
  The KM method will be used to summarize ADT-FS.
Time to progression | Time from completing SBRT to the time of first documented tumor progression or new lesions by PSMA PET/CT or initiation of ADT, assessed up to 60 months
Time to local progression (TTLP) | Time from completing SBRT to identification of progression of treated lesions, assessed up to 60 months
  The KM method will be used to summarize TTLP.
Time to new metastasis (TNM) | Time from completing SBRT to the time of a new documented tumor metastasis by PSMA PET/CT, assessed up to 24 months
  The KM method will be used to summarize TNM.
Overall survival (OS) | Time from starting treatment until death due to any cause, assessed up to 60 months
  The KM method will be used to summarize OS.
Local control (LC) | Time from starting treatment until local relapse is documented by PSMA PET/CT based criteria, assessed up to 24 months
  The KM method will be used to summarize LC.
Regional control (RC) | Time from starting treatment until regional relapse is documented by PSMA PET/CT based criteria, assessed up to 24 months
  failure in an adjacent lymph node region (for nodal targets) detected by PSMA PET/CT
Duration of complete response (CR) or partial response (PR) | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that current or progressive disease is objectively documented, assessed up to 60 months
  The KM method will be used to summarize the duration of complete or partial response.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Kishan AU, Valle LF, Wilhalme H, Felix C, Nabong R, Juarez-Casillas JE, Flores K, Ma TM, Ludwig V, Nakayama M, Ells Z, Dahlbom M, Lauria M, Meyer C, Cao M, Weidhaas JB, Telesca D, McGreevy K, Nickols NG, Karasik D, Parmisano S, Basehart TV, Brisbane W, Marks L, Rettig MB, Reiter RE, Boutros PC, Allen-Auerbach M, Czernin J, Steinberg ML, Calais J. 177Lu-Prostate-Specific Membrane Antigen Neoadjuvant to Stereotactic Ablative Radiotherapy for Oligorecurrent Prostate Cancer (LUNAR): An Open-Label, Randomized, Controlled, Phase II Study. J Clin Oncol. 2025 Dec 20;43(36):3812-3821. doi: 10.1200/JCO-25-01553. Epub 2025 Nov 12. PMID 41223345